CLINICAL TRIAL: NCT04404023
Title: A Phase I, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of a Single Dose of UB-221 in Healthy Volunteers
Brief Title: Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of UB-221 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UBP Greater China (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UBP-A124-IgE
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- UB-221 (0.2 mg/kg) (Experimental): Intravenous infusion
  Interventions: Biological: UB-221
- UB-221 (0.6 mg/kg) (Experimental): Intravenous infusion
  Interventions: Biological: UB-221
- UB-221 (2 mg/kg) (Experimental): Intravenous infusion
  Interventions: Biological: UB-221
- UB-221 (6 mg/kg) (Experimental): Intravenous infusion
  Interventions: Biological: UB-221
- UB-221 (10 mg/kg) (Experimental): Intravenous infusion
  Interventions: Biological: UB-221

INTERVENTIONS:
Biological: UB-221 — UB-221 (75 mg/ml)

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of a single dose of UB-221 in healthy volunteers.

DETAILED DESCRIPTION:
This is a phase I, open-label, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics,and immunogenicity of a single dose of UB-221 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with age between 20 to 65 years old (inclusive).
* Subjects who are able and willing to provide the informed consent.
* Male subjects with body weight of 50 kilogram (kg) or above; female subjects body weight of 45 kilogram (kg) or above.
* Researchers based on medical history, physical examination, vital signs, clinical laboratory results and 12-lead electrocardiogram identified healthy subjects without clinically significant abnormalities

Exclusion Criteria:

• The investigator considered that the subjects were not suitable to participate in this study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
1.Adverse event incidence | 15 days
  from the baseline to day 15 after IP infusion